CLINICAL TRIAL: NCT06802393
Title: Implementation of a Pharmacist-Led Social Determinants of Health Screening Intervention During Transitions of Care in an Acute Care Setting
Brief Title: Pharmacist-Led SDoH Screening Intervention During Transitions of Care in an Acute Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Matthew Jacobs, Associate Professor, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00007867; K23HL153582 (NIH)
Record Dates: First submitted 2025-01-23; First posted 2025-01-31 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-01

CONDITIONS: Health Related Social Needs (HRSN); Pharmacy; Medication Reconciliation
Keywords: health related social needs; pharmacists; hospital; emergency department; medication reconciliation
MeSH Terms: conditions — Emergencies | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The intervention study employs a quasi-experimental pre-post design with a non-equivalent control group to evaluate the impact of a pharmacist-led health-related social needs (HRSN) screening and referral intervention in an acute care setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention
  Interventions: Other: Intervention
- Control (Other): Control
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — The intervention incorporates a multifaceted pharmacist-led approach to addressing health-related social needs (HRSN) during transitions of care in the emergency department (ED) at Buffalo General Medical Center (BGMC). The intervention includes: 1) pharmacist-led medication reconciliation, and 2) HRSN screening using the Accountable Health Communities (AHC) HRSN tool. Based on the results, patients receive tailored referrals to community-based organizations using the 211 WNY database, which provides localized resources aligned with their social needs. Each patient is given a printed handout detailing the referral information. Within one month, a follow-up phone call is conducted to follow up with patients and assess additional needs as well as collect feedback through a patient satisfaction survey.
  Arms: Intervention
Other: Control — The control arm of the study consists of a historical cohort of patients who were admitted to or discharged from the emergency department (ED) at Buffalo General Medical Center (BGMC) during the same timeframe as the intervention arm but did not receive the pharmacist-led health-related social needs (HRSN) screening or referral intervention. These patients are identified through the electronic health record (EHR) based on the same inclusion criteria as the intervention group, such as age, geographic location, and discharge disposition. Control participants are matched 1:1 with intervention participants using demographic and clinical characteristics, including age (within 5 years), zip code, insurance type, discharge status, and race. Data for the control arm include healthcare utilization metrics such as 30- and 90-day unplanned hospital readmissions and emergency department visits. The control arm serves as a comparator to evaluate the effectiveness of the intervention
  Arms: Control

SUMMARY:
The study is a quasi-experimental pilot study conducted at Buffalo General Medical Center (BGMC). It aims to evaluate the feasibility, acceptability, and effectiveness of a pharmacist-led intervention addressing health-related social needs (HRSN) during transitions of care in the emergency department. The intervention involves: 1) pharmacist led medication review, 2) screening patients using the Accountable Health Communities (AHC) HRSN tool, connecting them to local community-based organizations, and 3) conducting follow-up to assess outcomes. The study will recruit 150 patients (50 intervention and 100 control) and assess healthcare utilization metrics, including hospital readmissions and emergency department visits.

DETAILED DESCRIPTION:
The study is a quasi-experimental pilot project conducted at Buffalo General Medical Center (BGMC). Using a pre-post design with a non-equivalent control group, the study aims to evaluate the feasibility, acceptability, and effectiveness of a pharmacist-led intervention addressing health-related social needs (HRSN) during care transitions in the emergency department (ED). Eligible patients, including English-speaking adults aged 18 or older will be identified daily through the ED worklist by trained research assistants. Participants will undergo screening using the Accountable Health Communities (AHC) HRSN tool to identify unmet needs such as housing instability, food insecurity, and transportation challenges.

The intervention includes: 1) pharmacist led medication reconciliation, 2) providing patients with tailored referrals to community-based organizations identified through the 211 WNY resource database, based on their specific social needs and geographic location and 3) follow-up phone calls within one month will assess whether participants contacted the referred organizations and whether these services were helpful. A patient satisfaction survey will also be conducted during these follow-up calls to gauge attitudes toward the intervention.

The historical control group will include patients admitted or discharged from the ED during the same timeframe as the intervention group but without HRSN screening. Control group data, including healthcare utilization outcomes, will be extracted from the electronic health record (EHR). Outcomes of interest include feasibility measures such as recruitment rates and data completeness, acceptability metrics like patient satisfaction, and secondary outcomes such as unplanned hospital readmissions and ED visits at 30 days and 3 months post-discharge.

Data analysis will involve statistical comparisons of demographic and clinical characteristics between the intervention and control groups using Chi-square tests for categorical variables and Wilcoxon Rank-sum or t-tests for continuous variables. Multivariable logistic regression will assess the impact of the intervention on healthcare utilization outcomes.

The study expects to recruit 50 patients in the intervention group and 100 in the control group over eight months, with a total study duration of 12 months, including follow-up and data analysis. By integrating pharmacists into HRSN screening and referral processes, the study aims to address critical social determinants of health, improve care transitions, and reduce healthcare utilization in underserved populations.

ELIGIBILITY:
Inclusion Criteria:

Age: Patients must be at least 18 years old.

Status: Patients being seen at Buffalo General Medical Center (BGMC).

Discharge Plan: It is anticipated that the patient will be discharged home. Control Group: Patients in the control group will meet the same inclusion criteria as those in the intervention group, except they will not receive the health-related social needs (HRSN) screening.

Exclusion Criteria:

Cognitive Impairment: Patients who are cognitively impaired and unable to consent will be excluded.

Non-English Speakers: Non-English speaking individuals are excluded due to the nature of the intervention requiring direct communication between the clinical pharmacist and participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Healthcare Utilization | 30 days post discharge
  The primary outcome measure of the study is the composite rate of unplanned, all-cause hospital readmissions or emergency department (ED) visits within 30 days of hospital discharge.

SECONDARY OUTCOMES:
Intervention feasibility and fidelity metrics | Through study completion and up to 30 day post discharge
  Recruitment Rates: The proportion of eligible patients who are approached and consented for the intervention.
  Completion Rates: The number of patients who complete all aspects of the intervention, including follow-up and patient satisfaction surveys.
  Follow-Up Rates: The proportion of participants who successfully engage with referred community-based organizations (CBOs).
Intervention Acceptability | Through study completion and up to 30 days post-discharge
  Patient satisfaction with the HRSN screening and referral process, assessed through post-intervention surveys.
  Participant attitudes toward pharmacist-led social care interventions in an acute care setting.
Rates of unplanned hospital readmissions and emergency department visits | Up to 90 days post-discharge
  Rate of Unplanned, All-Cause Hospital Readmissions at 30 and 90 Days: This evaluates the frequency of unplanned hospital readmissions within 30 and 90 days post-discharge in both the intervention and control groups.
  Rate of Unplanned, All-Cause Emergency Department (ED) Visits at 30 and 90 Days: This measures the number of unplanned ED visits within 30 and 90 days post-discharge for both groups, providing additional insights into healthcare utilization.

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo General Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No